CLINICAL TRIAL: NCT03749772
Title: Effectiveness of a Cognitive Training Therapy for Overweight/Obesity Treatment: A Randomized Clinical Trial.
Brief Title: Cognitive Therapy Plus Dietary Intervention for Obesity Treatment
Acronym: COGNI-OB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Juan Jose Hernández Morante, Professor, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PMAFI14/12-2
Record Dates: First submitted 2018-11-20; First posted 2018-11-21 (Actual); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Overweight and Obesity
Keywords: obesity, cognitive therapy, executive function
MeSH Terms: conditions — Overweight; Obesity | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Randomization was performed by the principal investigator. The interventions were carried out individually, so the participants were unaware of the existence of another study arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive (Experimental): The participants of the COGNITIVE group performed cognitive training during 12 sessions during the 3 months of hypocaloric treatment. The training was carried out with the PC game Brain Exercise TM (Bandai Namco Games Ltd.). The participants made a total of 12 practice exercises, which implies approximately 30 minutes of duration per session.
  Interventions: Behavioral: Cognitive Training
- Control (No Intervention): As a control group, we used nutrition education sessions of approximately the same duration (30 min) where we simply reinforced the knowledge that was already provided during the sessions with the patient, such as concepts about the balanced diet, nutrient composition and micronutrients, etc. The objective of this control group was to avoid the effect of time with the researcher.

INTERVENTIONS:
Behavioral: Cognitive Training — The intervention was carried out with the PC game Brain Exercise TM (Bandai Namco Games Ltd.). Participants held the training sessions on an HP 250 G3 Notebook PC (Windows 10), with a 15-inch screen, and a resolution of 1366x768x40 Hz. The performance achieved by each participant in each session was recorded to analyze the evolution of the subjects. The participants made a total of 12 practice exercises, which implies approximately 30 minutes of duration per session.
  Other Names: Cognitive Rehabilitation Therapy; Executive Function Training
  Arms: Cognitive

SUMMARY:
This randomized clinical trial was carried out from January 2017 to December 2017 at the facilities of the Catholic University of Murcia. Written informed consent was required from each patient. The protocols of the present clinical trial follow the CONSORT standards. To measure the impact of cognitive training on weight loss in overweight / obese subjects, a double-blind study (de facto masking) was designed.

Both the participants and the statistical assessors were unaware of the study hypothesis. Participants were unaware of treatments and possible assignments between groups, and only those subjects who were randomly assigned to the cognitive training group were informed that such training was part of dietary therapy.

The principal investigator of the present study (J.J.H.M.) carried out the randomization, with the assistance of the Microsoft Excell program, with the help of a macro designed in Visual Basic® for that purpose.

The randomization divided the subjects into two groups, as they were treated with a hypocaloric diet plus 12 nutrition education sessions (CONTROL group) or a group that were treated with a hypocaloric diet plus 12 sessions of cognitive training (COGNITIVE group).

In order to obtain a similar size in both groups, a randomization in blocks with a 1: 1 allocation ratio was performed.

Cognitive performance measures were performed before and after training. One week before the beginning of the cognitive and dietary intervention, the participants performed a series of cognitive tests. After 12 weeks of both dietary and cognitive intervention, participants were reexamined to measure performance on neurocognitive tests.

ELIGIBILITY:
Inclusion Criteria:

* Present a BMI> 27 kg / m2, and want to be part of the study voluntarily

Exclusion Criteria:

* subjects with diabetes mellitus type 2
* subjects with a history of a cardiovascular event (acute myocardial infarction, intermittent claudication, etc.)
* subjects with kidney or liver failure or some other significant pathology (cancer)
* subjects under pharmacological treatment that could affect body weight (corticoids, thyroxine, etc.)
* subjects who were on a diet or had been on a diet at least 6 months before their participation in the study were also excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2016-12-21 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Total weight loss percentage | 12 weeks
  Percentage of weight loss from baseline measurement to the end-of-treatment weight, calculated as (baseline weight - weight at week 12)/baseline weight * 100